CLINICAL TRIAL: NCT04459780
Title: Characterization and Functionality of Calcium Channels Cav1.4 of Th17 Lymphocytes in Human With Psoriasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Collaborators: Centre National de la Recherche Scientifique, France (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CaPSO17
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Psoriasis
Keywords: Th17; Cav1.4; Lymphocyte; Channel
MeSH Terms: conditions — Psoriasis; Cone-Rod Dystrophy, X-Linked, 3 | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Monocentric, open-label, comparative, parallel group and intra-individual patho-physiological study :
  * Group 1 : 20 subjects with plaque psoriasis
  * Group 2 : 10 subject with atopic dermatitis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 : 20 subjects with plaque psoriasis (Experimental): Intervention: skin biopsies and blood sample
  Interventions: Biological: Skin biopsies; Biological: Blood sample
- Group 2 : 10 subjects with atopic dermatitis (Experimental): Intervention: skin biopsies
  Interventions: Biological: Skin biopsies

INTERVENTIONS:
Biological: Skin biopsies — 3 biopsies on lesion skin (and one more for the first fifteen subjects in group 1)
Biological: Blood sample — One blood sample for the group 1 only.
  Arms: Group 1 : 20 subjects with plaque psoriasis

SUMMARY:
It's clearly known that lymphocyte activation in particular Th17 response, plays a major role in the development of plaque psoriasis. New therapies targeting this pathway are showing great clinical efficacy in patients with moderate to severe plaque psoriasis.

Pioneering observations have shown that the expression of Cav1.4 channels in Th17 lymphocytes and they're functional role is supported by the inhibition of IL-17 production by a pharmacological inhibitor of Cav1 channels that is effective in a mouse model of Psoriasis.

This data strongly suggest that the Cav1.4 channel, via its involvement in the signalling responsible for the production of Th17 cytokines represents an interesting therapeutic target in Psoriasis.

The aim of the study is to explore biological functions related to the activation of the Cav1.4 pathway in Psoriasis.

DETAILED DESCRIPTION:
* Evaluate the expression of Cav1.4 calcium channels by Th17 lymphocytes from plaque psoriasis.
* To assess:

  * The role of Cav1.4 channels on the activation of Th17 lymphocytes
  * The transcriptomic signature relating to the signalling channel Cav1.4
  * The epigenetic signature, in particular changes in overall methylation and specific promoter methylation

ELIGIBILITY:
Inclusion Criteria:

* Group 1 : Subject with plaque psoriasis (diagnosis confirmed by dermatologist) with a plaque IGA score ≥ 3
* Group 2 : Subject with atopic dermatitis according to the UK Working party criteria with an IGA plaque score ≥3

Exlusion Criteria:

* Group 1 : Other chronic inflammatory dermatosis than plaque psoriasis at the sites to be sampled
* Group 2 : Other chronic inflammatory dermatosis than Atopic Dermatitis at the sites to be sampled
* For both groups: Ongoing treatment with calcium channel blockers
* For both groups: Any current topical treatment on the biopsied or systemic plaque for psoriasis or AD (including phototherapy)

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-10-25 (Actual); Primary Completion 2017-11-13 (Actual); Study Completion 2017-11-13 (Actual)

PRIMARY OUTCOMES:
Expression of Cav1.4 calcium channels in Th17 lymphocytes | Baseline
  Immunohistochemistry (IHC) and in situ hybridation (HIS)

SECONDARY OUTCOMES:
Role of Cav1.4 channels on the activation of Th17 lymphocytes | Baseline
  Fonctional study : intracellular marquing and qPCR (with TLDA technology (TaqMan Low Density Arrrays)) and ELISA method
Transcriptomic signature relating to the signaling channel Cav1.4 | Baseline
  qPCR with TLDA technology (TaqMan Low Density Arrrays)
Epigenetic signature, in particular changes in overall methylation and specific promoter methylation | Baseline
  Pyrosequencing

CONTACTS AND LOCATIONS:
Overall Officials: Paul CARL, Pr., Principal Investigator — Service de Dermatologie - Hôpital Larrey
Locations (1):
- Service de Dermatologie - Hôpital Larrey, Toulouse, France

IPD SHARING:
Plan to Share IPD: No